CLINICAL TRIAL: NCT01659671
Title: RCT of the Effect of Uvulopalatopharyngoplasty Compared to Expectancy in Patients With Obstructive Sleep Apnea
Acronym: SKUP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Danielle Friberg, Associate Professor, MD, Senior Surgeon, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007/449-31/3, Ö 21-2007; 2007/449-31/3, Ö 21-2007 (Other: Ethic Committee, Karolinska Institutet, Stockholm, Sweden)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uvulopalatopharyngoplasty (Active Comparator): One arm is Uvulopalatopharyngoplasty(intervention group of 32 patients), one arm is expectancy (control group of 33 patients). After six months the controls have delayed surgery and then both groups are followed for two years
  Interventions: Procedure: Uvulopalatopharyngoplasty
- Control (Active Comparator): After six months the controls have delayed surgery then are followed for 2 year
  Interventions: Procedure: Uvulopalatopharyngoplasty

INTERVENTIONS:
Procedure: Uvulopalatopharyngoplasty — Uvulopalatopharyngoplasty: Resection of the soft palate 3 mm and tonsillectomy, amputation of the uvula to approx 1 cm, single sutures of the posterior pillar to the anterior pillar and of the soft palate.

SUMMARY:
Hypothesis:Pharyngeal surgery (UPPP) reduces significantly the nightly respiratory breathing pauses (apnoeas-hypopnoeas) and improves the daytime symptoms compared to expectancy for 6 months in patients with OSAS.

Background: Obstructive sleep apnea syndrome (OSAS) is associated with an increased risk of poor sleep quality, excessive daytime sleepiness and prolonged reaction time, which can elevate the risk for traffic accidents. Increased morbidity and three to four times increased mortality in these patients are well documented, mainly in the cardiovascular field. Pharyngeal surgery, i.e. uvulopalatopharyngoplasty (UPPP) opens up the airway and was the predominant treatment for OSAS worldwide before continuous positive airway pressure (CPAP) devices became widely available in the 1990s. Since then, the main treatment for OSAS has been CPAP, but an increasing number of patients are also treated with mandibular retaining device (MRD). UPPP as treatment for OSAS has been performed for 30 years. The evidence-grade for the efficacy has so far been very low, and the side-effects and complication rate has raised the question whether there is a place for surgical treatment of OSAS. However, the compliance for CPAP and dental devices are quite low (50-60%), leaving a lot of patients untreated if surgery is not offered. RCT UPPP is still missing and called for.

ELIGIBILITY:
Inclusion Criteria:

ApnéHypopnéIndex, AHI >14,9 Daytime sleepiness w Epworth sleepiness scale, ESS> 7 Sleepy during daytime 3-5 times per week or more BodyMassIndex, BMI < 36,0 Friedman staging system of tonsil size and tongue: i and II Patients w Friedman stage I and BMI < 30,0 could be directly included if patient positive and no contra-indications for surgery. All others should be failure of CPAP and MRD before inclusion.

Exclusion Criteria:

Other OSAS treatment during study, i.e., patient is clinically severely deteriorated.

Negative to surgery Night-shift worker Friedman stage III or IV Morbid obesity BMI >35,9 Severe psychological or neurological disease ASA class >3 Severe lung- or heart disease (not applicable for hypertension, nor stroke or MI more than after 2 years).

Insufficient knowledge in Swedish language (important for filling in questionnaires) Dangerous in traffic while driving Severe nasal congestion (can be included after successful treatment) Previous tonsillectomy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Changes in apnea-hypopnea index | 6 months and 2 years
  Apnea-hypopnea index (AHI) is the number of apneas or hypopneas per sleep hour. Polysomnography (PSG) is the Golden standard to use when measuring the AHI. PSG is the method we are using

SECONDARY OUTCOMES:
Changes in Epworth sleepiness scale | 6 months and 2 years
  Epworth sleepiness scale is a validated questionnaire. It consists of eight questions concerning the patients´ ability to fall asleep in different situations. The total sum is 24.

OTHER OUTCOMES:
Changes in Oxygen desaturation index | 6 months and 2 years
  Oxygen desaturation index (ODI) is the number of oxygen desaturations of 3 % or more per sleep hour.
changes in blood samples | 6 months 2 years
  Hb, LPK, CRP, cortisol, TSH, T4, ASAT, ALAT, ALP, γ-GT, CDT, Leptin/ghrelin, fB-Glucose, f-insulin, HDL, LDL, Cholesterol, Triglycerides, TNF-α, IL-1, IL-6
changes in score of SF 36 quality of life questionnaire | 6 months and 2 years
  QoL SF 36 validated questionnaire
changes in blood pressure | 6 months and 2 years
  systolic and diastolic morning pressure from arm
changes in vigilance | 6 months and 2 years
  modified Osler test
number of patients with serious complications from surgery | 6 months
number of patients with side-effects from surgery | 6 months and 2 years
  answers from a local questionnaire regaring pharyngeal side-effects
Changes in score of FOSQ questionnaire | 6 months and 2 years
  Validated questionnaire designed for patients with obstructive sleep apnea syndrome
identifying success factors for outcome of surgical intervention | 6 months 2 years
  Correlate for example tonsil size and tongue position (stageing system) with changes in AHI
changes in arousal index | 6 months and 2 years
  Polysomnographic results
changes in lowest oxygen saturation during sleep | 6 months 2 years
  Polysomnographic results
changes in ODI during REM sleep | 6 months 2 years
  Polysomnographic results
changes in ODI in supine position | 6 months 2 years
  Polysomnographic results
changes in time in supine position | 6 months and 2 years
  Polysomnographic results
changes in Body Mass Index | 6 months and 2 years
changes in RERA index | 6 months and 2 years
  Polysomnographic results, RERA are the respiratory effort related arousals during sleep
changes in mean length apneas and hypopneas | 6 months and 2 years
  Polysomnographic results
changes in AHI supine position | 6 months 2 years
  Polysomnographic results
changes in AHI in REM | 6 months and 2 years
  Polysomnographic results
changes in total sleep time | 6 months and 2 years
  Polysomnograåhic results
changes in RDI | 6 months and 2 years
  Polysomnographic results; RDI is the sum of AHI and RERA index

CONTACTS AND LOCATIONS:
Overall Officials: Danielle K Friberg, MD, PhD, Associate professor, Principal Investigator — Karolinska University Hospital, Karolinska Institutet
Locations (1):
- ORL dep, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Joar S, Danielle F, Johan B, Arne L, Roberta N, Nanna B. Sleep Quality After Modified Uvulopalatopharyngoplasty: Results From the SKUP3 Randomized Controlled Trial. Sleep. 2018 Jan 1;41(1). doi: 10.1093/sleep/zsx180. PMID 29099950
- [Derived] Fehrm J, Friberg D, Bring J, Browaldh N. Blood pressure after modified uvulopalatopharyngoplasty: results from the SKUP3 randomized controlled trial. Sleep Med. 2017 Jun;34:156-161. doi: 10.1016/j.sleep.2017.02.030. Epub 2017 Apr 4. PMID 28522085
- [Derived] Browaldh N, Bring J, Friberg D. SKUP(3) RCT; continuous study: Changes in sleepiness and quality of life after modified UPPP. Laryngoscope. 2016 Jun;126(6):1484-91. doi: 10.1002/lary.25642. Epub 2015 Sep 25. PMID 26404729
- [Derived] Browaldh N, Nerfeldt P, Lysdahl M, Bring J, Friberg D. SKUP3 randomised controlled trial: polysomnographic results after uvulopalatopharyngoplasty in selected patients with obstructive sleep apnoea. Thorax. 2013 Sep;68(9):846-53. doi: 10.1136/thoraxjnl-2012-202610. Epub 2013 May 5. PMID 23644225